CLINICAL TRIAL: NCT00595088
Title: Phase 2b, Multicenter Trial of Intravesical DTA-H19/PEI in Patients With Intermediate-Risk Superficial Bladder Cancer
Brief Title: Phase 2b, Trial of Intravesical DTA-H19/PEI in Patients With Intermediate-Risk Superficial Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anchiano Therapeutics Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-07-01.CTIL
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2013-08-21 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Superficial Bladder Cancer
Keywords: Bladder Cancer; Refractory; inodiftagene vixteplasmid
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 20 mg of BC-819/PEI (Experimental): Six intravesical instillations of 20 mg of plasmid DNA (BC-819) complexed with PEI into the bladder of patients with intermediate-risk superficial bladder cancer [recurrent stages Ta (low or high grade) and T1 (low grade) TCC] who have failed prior intravesical therapies including BCG and/or chemotherapy.
  Interventions: Biological: BC-819/PEI

INTERVENTIONS:
Biological: BC-819/PEI — Papillary tumors will be resected with the exception of one marker tumor that will remain to examine the effects of the treatment on the remaining tumor. Study treatments will consist of an induction course of six weekly instillations of 20 mg of DTA-H19/PEI into the urinary bladder. Intravesical therapy will be delivered through a Foley catheter. Patients will be instructed to hold the dose in the bladder for two hours after administration. If the patient has a complete response, then she/he will be eligible to receive three additional courses of 3 weekly intravesical administrations of the same dose of investigational product every 12 weeks.
  Other Names: DTA-H19

SUMMARY:
This study is designed to assess the efficacy and safety of DTA-H19/PEI given as six intravesical instillations of 20 mg of plasmid DNA complexed with PEI into the bladder of patients with intermediate risk superficial bladder cancer [recurrent stages Ta (low or high grade)and T1, (low grade) transitional cell carcinoma (TCC)] who have failed prior intravesical therapies including either Bacillus Calmette-Guérin (BCG) or chemotherapy. The primary efficacy objective is to determine the effect of DTA-H19/PEI on the prevention of new tumors after the induction course of 6 weekly intravesical administrations of investigational product assessed 8 to 10 weeks after the start of treatment. Secondary objectives include assessing the ablative effect of DTA-H19/PEI on a marker tumor, safety assessed by the incidence and severity of adverse events, determining the long-term (46 weeks) continued rates of absence of bladder cancer, and time to tumor recurrence in those patients who had a complete response (CR) after the induction course.

DETAILED DESCRIPTION:
DTA-H19, is a doubled stranded DNA plasmid that carries the gene for the diphtheria toxin A (DT-A) chain under the regulation of the H19 promoter sequence. This is a Patient-Oriented, Targeted Therapy as DT-A chain expression is triggered by the presence of H19 transcription factors that are upregulated in tumor cells. The selective initiation of toxin expression results in selective tumor cell destruction via inhibition of protein synthesis in the tumor cell, enabling highly targeted cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, patients must:

1. Provide written informed consent.
2. Have intermediate-risk recurrent superficial TCC of the bladder defined as Stage Ta (low or high grade) or T1 (but with penetration into no more than ½ of the lamina propria), low grade (grade 1 or grade 2), as confirmed by histopathology, and have not recurred within 3-months of a complete course of a prior acceptable therapy (i.e., 6-weekly intravesical administrations of BCG or standard adjuvant treatment with thiotepa, doxorubicin, epirubicin, valrubicin, or mitomycin C).
3. Have complete resection of all papillary tumors with the exception of a single superficial papillary tumor that is appropriate to be a marker tumor (<1 cm in diameter).
4. Have ≥ 2 tumor and ≤ 7 tumors visible during cystoscopy and no tumor larger than 3 cm in diameter. If only one tumor is present, it must be large enough to obtain a biopsy specimen adequate to determine the tumor stage and grade and leave a marker tumor.
5. Have at least one tumor specimen resected before the start of the study that was positive for H19 expression by ISH. H19 expression positive is defined as >= 60 % of the tumor cells in the specimen expressing H19 at a moderate staining intensity.
6. Have failed at least one prior standard intravesical treatment including chemotherapy with mitomycin C, thiotepa, valrubicin, doxyrubicin, or epirubicin, or immunotherapy with BCG. Failure after treatment with chemotherapy is defined as recurrent disease after at least one intravesical instillation of drug. Failure after treatment with BCG is defined as intolerance to treatment such that treatment was discontinued or after having received 6 or more BCG instillations there is recurrent or persistent disease 3 or more months after initiation of BCG treatment.
7. Have a Karnofsky's performance status of greater than or equal to 60%.
8. Have adequate bone marrow reserve: Hemoglobin > 10 g/dL, WBC greater than or equal to 3000/mm3, and platelets > 100,000 /mm3.
9. Have adequate renal function with serum creatinine < 1.5 x the laboratory upper limit of normal (ULN).
10. Have adequate liver function with serum biliru¬bin, AST/SGOT and ALT/SGPT < 2 times the laboratory ULN.
11. Be at least 18 years of age.
12. If male, agree to use a condom, if sexually active, and if female, agree to practice one of the acceptable methods of birth control or be surgically sterile or postmenopausal (greater than 1 year post last menstrual cycle.

Exclusion Criteria:

To be eligible to participate in this study, patients must not:

1. Have current diagnosis or history of Stage T1 (high grade) or Stage T2 or higher or CIS.
2. Have severe concomitant disease that might limit compliance or completion of the protocol.
3. Have a tumor in a diverticulum, in the prostatic urethra, or covering the ureteral orifice.
4. Have any other malignancy that might impact 5-year survival or might be potentially confused with TCC.
5. Have congenital or acquired immune deficiencies.
6. Be receiving cytotoxic drugs or corticosteroids.
7. Have received intravesical therapy within 8 weeks prior to study entry.
8. Have received radiation therapy for their bladder cancer at any time or any other conditions including pelvic irradiation for any condition within 4 months prior to study entry.
9. Have active infections (including urinary tract infections) defined as viral, bacterial, or fungal infections requiring therapy, HIV-positive status, concurrent febrile illness, or gross hematuria.
10. Have biopsy, TUR, or traumatic catheterization within 14 days of start of treatment.
11. If female, be pregnant or breast feeding.
12. Have participated in any therapeutic research study within the last 8 weeks.
13. Have participated in any other gene therapy study including patients who have received DTA-H19/PEI in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Lamm, MD, Principal Investigator — University of Arizona and BCG Oncolgy
Locations (6):
- BCG Oncology, Phoenix, Arizona, United States
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah and Hebrew University Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Assaf Harofeh, Zrifin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit 12 Feb 2008, Last patient first visit 19 Sep 2012. All patients were recruited at the medical sites
Pre-assignment Details: Patients had to be H19 positive to be recruited
Period: Overall Study
Arm/Group | 20 mg of BC-819/PEI
Started | 47
Completed | 7 (5 patients ongoing, 7 completed the study (week 46)and 35 withdrew prematurely)
Not Completed | 40

BASELINE CHARACTERISTICS:
Arm/Group | 20 mg of BC-819/PEI
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 31
Sex: Female, Male [Count of Participants; unit: Participants] — 36 males and 11 females
  Participants
    Female | 11
    Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 8
  Israel | 39

OUTCOME MEASURES:

1. Primary Outcome: Complete Tumor Response Defined as the Absence of New Tumors
Description: Tumor response evaluated at week 9 (range 8-10 weeks) during the first post induction course treatment cystoscopy or TUR of suspiciaous lesions
Time Frame: 9 Weeks
Population: All patients who met the study inclusion and exclusion criteria; received all 6 of the induction course intravesical administrations of the investigational product; and had a follow-up cystoscopy during Weeks 8 to 10 and biopsy or TUR of suspicious lesions
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | 20 mg of BC-819/PEI
Number analyzed (Participants) | 39
percentage of participants | 64.1 [49.7 to 76.8]

2. Secondary Outcome: Time to Tumor Recurrence
Description: The Time to Tumor Recurrence is defined as the interval between the date of the final tumor resection before the start of study treatments to the date when the cystoscopy was performed in which it was confirmed by histopathology that any suspicious lesions that were observed, were TCC of the bladder with the exception of the continued presence of the marker tumor at Week 9
Time Frame: 46 Weeks
Measure: Median (Full Range); unit: months
Arm/Group | 20 mg of BC-819/PEI
Number analyzed (Participants) | 39
months | 11.3 [2.4 to 52.2]

3. Secondary Outcome: Ablative Effect on a Marker Tumor
Description: Complete disappearance of marker lesion
Time Frame: 9 weeks
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | 20 mg of BC-819/PEI
Number analyzed (Participants) | 39
percentage of participants | 33.3 [21.0 to 47.7]

ADVERSE EVENTS:
Time Frame: Screening through Week 46
Arm/Group | 20 mg of BC-819/PEI
Serious Adverse Events (participants affected / at risk) | 3/47
Other Adverse Events (participants affected / at risk) | 35/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg of BC-819/PEI (N=47)
Urinary retention (Renal and urinary disorders) | 1 (1) — Hospitalization due to a urinary tract infection caused by urinary tract outlet obstruction associated with benign prostate hypertrophy. Treatment:indwelling catheter and one week of parenteral antibiotics
Transurethral prostactectomy (Renal and urinary disorders) | 1 (1) — Hospitalization for prostactectomy
Urinary tract infection (Renal and urinary disorders) | 1 (1) — UTI following urinary retention
Myocardial infarction (Cardiac disorders) | 1 (1) — Hospitalization for cardiac catheterization
Hematuria (Renal and urinary disorders) | 1 (1) — Hospitalization due to clot retention and macroscopic hematuria
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 20 mg of BC-819/PEI (N=47)
Nausea (Gastrointestinal disorders) | 3 (3)
Asthenia (General disorders) | 3 (9)
Chills (General disorders) | 3 (5)
Pyrexia (General disorders) | 3 (3)
Urinary tract infection (Renal and urinary disorders) | 5 (6)
Increased blood potassium (Infections and infestations) | 5 (7)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (3)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 6 (6)
Nervous system disorders (Nervous system disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 5 (18)
Micturition urgency (Renal and urinary disorders) | 3 (9)
Pollakiuria (Renal and urinary disorders) | 7 (12)
Urinary retention (Renal and urinary disorders) | 3/4 (3)
Respiratory and thoracic disorders (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No